CLINICAL TRIAL: NCT05783583
Title: A Comparison of the Diagnostic Confidence and Image Quality Between the Eyoto Theia (RDSL) Remote Digital Slit Lamp and a the Topcon SL-D2 With DC-4 Digital Attachment (Predicate Device).
Brief Title: A Comparison of the Diagnostic Confidence and Image Quality Between the Eyoto Theia (RDSL) and a Predicate Device.
Status: Completed | Type: Observational
Sponsor: Eyoto Group Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EYO-CS-001.1
Record Dates: First submitted 2023-01-30; First posted 2023-03-24 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Enrolled participants: Adult human subjects showing either healthy eyes or specific ocular pathologies.
  Interventions: Device: Remote Digital Slit Lamp

INTERVENTIONS:
Device: Remote Digital Slit Lamp — Slit Lamp Examination

SUMMARY:
A clinical study has been identified as a requirement for the RDSL (Theia). This study involves a clinical comparison of the imaging from the RDSL with that of a predicate device.

The clinical evaluation showed that there remains some residual risk in the practitioner's ability to use the imaging from the RDSL to detect pathologies at the same level as when using the imaging function on a predicate device.

The aim of this comparative study is to determine the degree, if any, of difference in using images captured from the RDSL for clinical inspection of pathologies, when compared to images captured from a predicate device.

Due to the involvement of real patients during the study, ethics approval was sought prior to commencement. This study is limited to the clinical benefits of the device.

An additional Human factors study has been conducted to assess the useability of the device Images were taken of healthy eyes and eyes with pathology (with images of several pathologies from each major pathology group to give a full range) on both the predicate device, and the RDSL.

DETAILED DESCRIPTION:
Methodology

Overview Images were taken of 14 healthy eyes and 35 unhealthy eyes containing a range of pathologies on both the predicate device and the THEIA. The pathologies to be imaged have been carefully selected using data from the clinical evaluation, and further investigation, to ensure that all aspects of the imaging systems and ocular structures are included.

The images were taken on compliant patients in a real-world setting.

Device Selection Device Type:AC-powered remote enabled slit-lamp Manufacturer:Eyoto Product Number:THEIA (3-008-0001-03)

Intended Use:

The THEIA is intended for non-invasive examination, illumination, magnification, visualization and recording of digital photographs and video of the anterior and posterior eye segments of the human eye and its surrounding area.

Magnification:6 (base Magnification), 10X, 16X, 25X (digital steps) Filters:Blue filter,Red-free filter (digital filter),yellow Filter (fluorescein enhancement filter) Lighting:White LED,12 V, 0.7 - 1.5 A, 8.4 W Image Sensor,CMOS, 1.1", 12 Megapixel The latest pre-production version of the THEIA was used. This is representative of and has all the same functionality as, the production model.

Three individual THEIA devices of the same version were used to collect the images.

Predicate Device Device Type:AC-powered slit lamp biomicroscope Manufacturer:Topcon Product Number:Topcon SL-2G or equivalent (SL-2D with imaging attachment) Intended Use:The Slit Lamp SL-2G is an AC-powered slit lamp biomicroscope intended for use in eye examination of the anterior eye segment, from the cornea epithelium to the posterior capsule. It is used to aid in the diagnosis of diseases or trauma which affect the structural properties of the anterior eye segment.

Magnification:10X, 16X, 25X Filters:Blue filter, Red-free filter, Yellow Filter (fluorescein enhancement filter) available as an accessory Lighting:White LED Image Sensor (DC-4):CMOS, 5 Megapixel

The predicate device used for this study was equivalent to the Topcon SL-2G used in the substantial equivalence investigation, used with the recommended Topcon Digital Imaging Adaptor (DC-4) in order to take the images required.

Three individual predicate devices will be used to collect the images.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eye or ocular pathology

Exclusion Criteria:

* No exclusion other than age as above

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic Confidence | Within 1 week after data collection
  How confident the practitioner is in respect of their identification of a pathology from image on a scale of 1-5, with 5 being completely confident and 1 being not confident. Images reviewed via online from.
Image Clarity | Within 1 week after data collection
  The rating of clarity of image by the practitioner on a scale of 1-5, with 5 being excellent clarity and 1 being low clarity. Images reviewed via online from.
Identification of Pathology | Within 1 week after data collection
  % accuracy of identification of pathology shown or healthy eye. Images reviewed via online from.

CONTACTS AND LOCATIONS:
Overall Officials: John Bankowski, DOO, Principal Investigator — National Vision Inc
Locations (1):
- National Vision Inc Corporate Office, Atlanta, Georgia, United States